CLINICAL TRIAL: NCT04645550
Title: Efficacy and Safety of Apixaban, Warfarin and Aspirin Anticoagulation for Prevention of Portal Vein Thrombosis in Liver Cirrhotic Patients After Laparoscopic Splenectomy
Brief Title: Apixaban, Warfarin and Aspirin Prevents Portal Vein Thrombosis in Patients After Laparoscopic Splenectomy（ESAWAAPT）
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, PhD, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YZUC-005
Record Dates: First submitted 2020-11-22; First posted 2020-11-27 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cirrhosis; Splenectomy; Status; Venous Thrombosis; Hypertension, Portal
Keywords: Cirrhosis; Venous thrombosis; Portal Hypertension; Apixaban; Warfarin; Aspirin; Splenectomy; Laparoscopy
MeSH Terms: conditions — Fibrosis; Venous Thrombosis; Hypertension, Portal | interventions — apixaban; Warfarin; Aspirin; aspirin, magnesium oxide combination; Dipyridamole; Heparin, Low-Molecular-Weight; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apixaban with dipyridamole (Experimental): From postoperative day 3, patients will receive oral dipyridamole 25mg tid for three months along with subcutaneous injection of Low Molecular Weight Heparin (4100 IU) for first five days and Apixaban 2.5mg bid for six months.
  Interventions: Drug: Apixaban; Drug: Dipyridamole; Drug: Low molecular weight heparin
- Warfarin with dipyridamole (Experimental): From postoperative day 3, patients will receive dipyridamole 25mg tid for three months along with subcutaneous Low Molecular Weight Heparin Calcium injection for first five days and Warfarin 2.5mg qd with titration of dose to maintain a target INR of 2-3. Intially the INR will be monitored twice weekly with gradual escalation of dose to achieve target INR. After achieving the target INR, this is to be repeated every 4 weeks. The Doppler Ultra Sonography screening will be done every 3 months to assess the occurrence of portal vein thrombus, but the medications will be continue for six months irrespective of the occurrence of portal vein thrombus.
  Interventions: Drug: Warfarin; Drug: Dipyridamole; Drug: Low molecular weight heparin
- Aspirin with dipyridamole (Experimental): From postoperative day 3, patients will receive oral dipyridamole 25mg tid for three months along with subcutaneous injection of Low Molecular Weight Heparin (4100 IU) for first five days and Aspirin Enterie Ccoated Tablets 100mg qd for six months.
  Interventions: Drug: Aspirin; Drug: Dipyridamole; Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Apixaban — From postoperative day 3, patients will receive oral Apixaban 2.5mg bid for six months.
  Other Names: ELIQUIS
  Arms: Apixaban with dipyridamole
Drug: Warfarin — From postoperative day 3, patients will receive oral Warfarin 2.5mg qd with titration of dose to maintain a target INR of 2-3 for six months.
  Other Names: Warfarin Sodium; Athrombine; COUMADIN; PANAWARFIN
  Arms: Warfarin with dipyridamole
Drug: Aspirin — From postoperative day 3, patients will receive oral Aspirin Enterie Ccoated Tablets 100mg qd for six months.
  Other Names: Acenterine; Acetard; Acetophen
  Arms: Aspirin with dipyridamole
Drug: Dipyridamole — From postoperative day 3, patients will receive oral dipyridamole 25mg tid for three months.
  Other Names: Gardoxin; Coribon; Curantyl; Dilaplus
Drug: Low molecular weight heparin — From postoperative day 3, patients will receive subcutaneous injection of Low Molecular Weight Heparin (4100 IU) once daily for first five days.
  Other Names: Fraxiparine

SUMMARY:
The purpose of this study is to determine whether Apixaban, Warfarin and Aspirin Anticoagulation are effective and safe in Prevention of Portal Vein Thrombosis in Liver Cirrhotic Patients after Laparoscopic Splenectomy

DETAILED DESCRIPTION:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have no portal vein thrombosis will be enrolled. The baseline Doppler parameter will be recorded and the patient will be randomized into apixaban, warfarin or aspirin group. From postoperative day three, patients in apixaban group will receive oral Apixaban 2.5mg bid for six months, patients in warfarin group will receive oral Warfarin 2.5mg qd with titration of dose to maintain a target INR of 2-3 for six months, patients in aspirin group will receive oral Aspirin Enterie Ccoated Tablets 100mg qd for six months. All groups will be along with five days of subcutaneous injection of Low Molecular Weight Heparin and three months of oral Dipyridamole. Every three months the Doppler screening for the occurrence of portal vein thrombus (PVT) or spleno-mesenteric thrombosis will be done for all patients. All groups will receive the therapy for six months irrespective of the Doppler findings in relation to portal vein thrombus occurrence. Then six months monitoring will be done in the three groups as per the primary or secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
* Splenomegaly with secondary hypersplenism
* No evidence of PVT or spleno-mesenteric thrombosis by ultrasound evaluation and angio-CT
* Informed consent to participate in the study

Exclusion Criteria:

* Hepatocellular carcinoma or any other malignancy
* Hypercoagulable state other than the liver disease related
* DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs
* Base line INR >2
* Child-Pugh grade C
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy
* Uncontrolled Hypertension
* Human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Proportions of patients who will suffer PVT or spleno-mesenteric thrombosis among oral anticoagulant Apixaban with dipyridamole group, oral Warfarin with dipyridamole group and oral Aspirin with dipyridamole group during the study period | Two years

SECONDARY OUTCOMES:
Proportions of patients who will show improvement in Child Pugh (>2 points) in three groups | Two years
Proportions of patients who will show improvement in Model for End Stage Liver Disease (MELD)(>4 points) in three groups | Two years
Proportions of patients who will show decrease in hepatic decompensation defined as development of ascites, PSE, portal hypertensive bleeding, jaundice, spontaneous bacterial peritonitis, or systemic infection | Two years
Proportions of patients who will suffer from hepatocellular carcinoma in three groups. | Two years
Overall survival in three groups. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Dou-Sheng Bai Bai, MD, Study Chair — Clinical Medical College of Yangzhou University; Guo-Qing Jiang, MD, Study Director — Clinical Medical College of Yangzhou University; Sheng-Jie Jin, MD, Principal Investigator — Clinical Medical College of Yangzhou University; Bao-Huan Zhou, MS, Principal Investigator — Clinical Medical College of Yangzhou University; Tian-Ming Gao, MS, Principal Investigator — Clinical Medical College of Yangzhou University
Locations (1):
- Clinical Medical College of Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No